CLINICAL TRIAL: NCT04686435
Title: Metabolic Syndrome and Persistent Shoulder Pain 1 Year After Primary Diagnosis: The Prospective Vejle Hospital Shoulder Cohort (VHS Cohort) With Focus on Prognostic Factors
Brief Title: Metabolic Syndrome and Persistent Shoulder Pain 1 Year After Primary Diagnosis
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Collaborators: Region of Southern Denmark (Other); The A.P. Moller Foundation (Unknown); The Lillebaelt Hospital Research Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: VHS Cohort 20/12316
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Pain; Metabolic Syndrome
MeSH Terms: conditions — Shoulder Pain; Metabolic Syndrome | interventions — Physical Therapy Modalities; Exercise; Adrenal Cortex Hormones; Dosage Forms; Acupuncture Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-surgical treatment: Shoulder patients referred for non-surgical treatment after being diagnosed at the medical examination.
  Interventions: Other: Non-surgical treatment such as physiotherapy, exercise, corticosteroid injection, medication, acupuncture
- Surgical treatment: Shoulder patients referred for surgical treatment after being diagnosed at the medical examination.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Other: Non-surgical treatment such as physiotherapy, exercise, corticosteroid injection, medication, acupuncture — Treatment consisting of different non-surgical interventions as recommended by the orthopedic specialist and decided upon in shared decision making with the patient
  Other Names: Physiotherapy; Exercise; Corticosteroid injection; Medication; Acupuncture
  Groups: Non-surgical treatment
Procedure: Surgery — Surgery can consist of rotator cuff repair, Bankart repair, subacromial decompression, biceps tenodesis or tenotomy, acromioclavicular joint resection.
  Groups: Surgical treatment

SUMMARY:
In a longitudinal cohort project, the objective is to evaluate general prognostic and individual risk factors for long lasting shoulder pain, with a specific focus on evaluation of the association between metabolic syndrome and tendinopathy, while simultaneous adjusting for other potential prognostic candidate variables (PROGRESS Theme I-II).

DETAILED DESCRIPTION:
The VHS Cohort is a prospective cohort trial evaluating a wide range of patient reported and clinical prognostic factors, attained prior to initiation of treatment, among shoulder patients referred for diagnostic evaluation at the specialized shoulder unit at Vejle Hospital, Denmark. The department receives approximately 2000 new patients each year.

Prior to medical examination, patients will be asked to fill in a baseline questionnaire, and from the electronic patient record, a range of different clinical factors will be obtained.

Subsequently, patients will be asked to answer questionnaires on patient reported outcomes after 1, 3, 6, and 12 months. Five years after inclusion into the trial, work affiliation will be retrieved from registries in order to evaluate association between shoulder disorders and work affiliation.

The objective of the VHS Cohort Project is to evaluate general prognostic and individual risk factors for long lasting shoulder pain. A specific focus is evaluation of the association between metabolic syndrome and rotator cuff tendinopathy while simultaneously adjusting for other potential prognostic candidate variables (PROGRESS Theme I-II). In a subsequent cohort (VHS Cohort Project II), the objective will be to develop a prognostic model for the treatment effect of Rotator Cuff Related Shoulder Pain (RCRSP) (PROGRESS Theme III).

VHS Cohort Project I:

Aim 1: Evaluate the risk of consistent pain one year after diagnosis among patients diagnosed with: RCRSP; Rotator cuff lesions (conservatively treated); Acromioclavicular osteoarthritis and Adhesive capsulitis (PROGRESS Theme I).

Aim 2: Evaluate the risk of consistent pain one year after surgery for: subacromial Decompression OR Rotator Cuff lesion (PROGRESS Theme I).

Aim 3: Evaluate the risk of consistent pain one year after diagnosis in patients with metabolic syndrome compared to patients without metabolic syndrome, with particular emphasis on patients diagnosed with RCRSP while simultaneously adjusting for other potential prognostic candidate variables (PROGRESS Theme II).

We hypothesize that

* Significantly more patients with RCRSP have metabolic syndrome than patients diagnosed with other shoulder-specific diagnoses
* Significantly more patients with metabolic syndrome and diagnosed with RCRSP are classified as non-responders to treatment than patients with other shoulder specific diagnoses 52 weeks after initial medical examination.
* Significantly more shoulder patients with metabolic syndrome report multiple musculoskeletal pain sites than shoulder patients without metabolic syndrome at first medical examination.

Aim 4: From clinical examination findings and patient reported information identify the strongest individual predictors of prognostic value for persistent shoulder pain and disability one year after initial medical examination in patients with rotator cuff related pain syndrome (RCRSP) (Diagnostic codes: DM75.1; DM75.1A; DM75.1B; DM75.4; DM75.5; DM75.8; DM75.9) treated conservatively with either exercise, corticosteroid injection, or a combination of the two, while simultaneously adjusting for other potential prognostic candidate variables (PROGRESS Theme II).

Aim 5: From clinical examination findings and patient reported information identify the strongest individual preoperative predictors of prognostic value for persistent shoulder pain and disability one year after surgery for patients receiving SubAcromial Decompression (SAD) surgery (Procedure code: KNBH51), while simultaneous adjusting for other potential prognostic candidate variables (PROGRESS Theme II).

Aim 6: From clinical examination findings and patient reported information, identify the strongest individual predictors of five-year work participation rates.

ELIGIBILITY:
Inclusion Criteria:

* Referred for medical examination to the shoulder sector, orthopedic Department, Vejle Hospital - Hospital Lillebaelt
* Older than 18 years
* Diagnosed with shoulder disorder at medical examination.

Exclusion Criteria:

* Significant cognitive impairment or language issues
* Symptomatic cervical spine pathology
* Older than 75 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will include all patients diagnosed with a shoulder disorder at their medical examination, and have given written consent to participate.
Sampling Method: Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with more than 41% improvement in disability 12 months after diagnosis as measured by Quick-DASH. | 12 months
  Quick-DASH (Disabilities of the Arm, Shoulder and Hand) is a patient reported questionnaire measuring upper extremity function and pain.

SECONDARY OUTCOMES:
Number of patients in the normal able-bodied population changing from "Being associated with the labour market" to "Not being associated with the labour market" in work participation classification. | 5 years
  Registry obtained information about participants work affiliation from diagnosis to five years after inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Kim G. Ingwersen, PhD, Principal Investigator — Vejle Hospital, University Hospital of Southern Denmark
Locations (1):
- Vejle Hospital, University Hospital of Southern Denmark, Vejle, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be shared upon direct contact to principal investigator with relevant purpose.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-08-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT04686435/SAP_000.pdf